CLINICAL TRIAL: NCT00707226
Title: Circadian Variations in Ocular Blood Flow in Glaucomatous and Normal Eyes
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Michael Georgopoulos, Medical University of Vienna
Other Study IDs: OPHT-171000
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2008-06-30 (Estimated); Status verified 2008-06

CONDITIONS: Glaucoma, Open-Angle; Circadian Rhythm; Intraocular Pressure; Regional Blood Flow
Keywords: Laser Doppler flowmetry; Choroidal blood flow; Fundus pulsation amplitude; Intraocular Pressure
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: 15 patients with primary open angle glaucoma
- 2: 15 age matched healthy subjects

SUMMARY:
After focusing many years only on intraocular pressure (IOP) as the primary risk factor, recently the impact of ocular blood flow is getting more consideration for the pathophysiology of glaucoma. The circadian change of intraocular pressure (IOP) is well investigated, but diurnal variations in ocular blood flow are yet to be evaluated, especially in glaucomatous eyes.

This study is performed to investigate circadian variation of ocular blood flow assessed by laser interferometric fundus pulsation amplitude (FPA) and laser Doppler flowmetry (LDF) in glaucomatous eyes during topical antiglaucoma therapy at 8:00, 12:00, 17:00 and 21:00, to compare these circadian variation of ocular blood flow in glaucomatous eyes with variations in healthy eyes and to relate blood flow variations with IOP variations.

ELIGIBILITY:
Inclusion Criteria:

For the glaucoma patients:

* Medical controlled Primary Open Angle Glaucoma with a history of more than 2 years
* Topical medication with beta-blockers (timolol, betaxolol, levobunol)
* IOP with medication < 22 mmHg (with a medical history of IOP > 22 mmHg)
* Visual field testing: mild glaucomatous defects (Humphrey 30-2 with MD>10)
* Optic nerve head: C/D-ratio between 0.4 and 0.9
* ametropy < 3 dpt
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

For the age matched control subjects:

* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 dpt.

Exclusion Criteria:

For the glaucoma patients:

* History of trabeculectomy or laser trabeculoplasty
* Any other ocular disease with possible vascular involvement such as diabetic retinopathy, age related macular disease, retinal vein or artery occlusion.
* Uncontrolled systemic hypertension (defined as systolic blood pressure > 170 mmHg or diastolic blood pressure > 100 mmHg)
* Diabetes mellitus

For the age matched control subjects:

* abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease
* Ametropy > 3 dpt

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-11; Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
fundus pulsation amplitude choroidal blood flow IOP | 13 hours

SECONDARY OUTCOMES:
blood pressure, pulse rate | 13 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Georgopoulos, MD, Principal Investigator — Department of Clinical Ophthalmology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria